CLINICAL TRIAL: NCT03503344
Title: A Randomized, Phase II Study of Apalutamide +/- Stereotactic Body Radiotherapy (SBRT) in Castration-Resistant Prostate Cancer Patients With Oligometastatic Disease on PSMA-PET Imaging
Brief Title: Apalutamide With or Without Stereotactic Body Radiation in Treating Castration-Resistant Prostate Cancer
Acronym: PILLAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Rahul Aggarwal, Associate Clinical Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 175519; NCI-2018-00572 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; PSA Progression; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — apalutamide; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (apalutamide monotherapy) (Experimental): Participants receive apalutamide PO QD on days 1-28. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Apalutamide
- Arm B (apalutamide, SBRT) (Experimental): Participants receive apalutamide PO QD on days 1-28. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Beginning 60 days after first dose of apalutamide, participants also undergo stereotactic body radiation therapy for 1-5 fractions.
  Interventions: Drug: Apalutamide; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Apalutamide — Given PO, 240 mg per day (4 x 60mg tablets)
  Other Names: ARN 509; JNJ 56021927
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm B (apalutamide, SBRT)

SUMMARY:
This phase II trial studies the how well apalutamide with or without stereotactic body radiation therapy work in treating participants with castration-resistant prostate cancer. Testosterone can cause the growth of prostate cancer cells. Hormone therapy using apalutamide may fight prostate cancer by blocking the use of testosterone by the tumor cells. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. It is not yet known whether giving apalutamide with or without stereotactic body radiation therapy works better in treating participants with castration-resistant cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate whether the proportion of patients with an undetectable serum prostate specific antigen (PSA) at 6 months following cessation of apalutamide is higher with addition of stereotactic body radiation therapy (SBRT) to prostate specific membrane antigen (PSMA)-avid oligometastatic sites of disease compared to the group of patients receiving apalutamide monotherapy

SECONDARY OBJECTIVES:

I. To compare the time to PSA progression by Prostate Cancer Working Group (PCWG) criteria between treatment arms.

II. To evaluate the safety and tolerability of apalutamide in combination with SBRT.

EXPLORATORY OBJECTIVES:

I. To characterize the metastatic pattern at baseline and at progression in these patients and to determine whether features of the baseline PSMA-PET scan are associated with treatment outcomes.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Participants receive apalutamide PO QD on days 1-28. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Participants receive apalutamide orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Beginning 60 days after first dose of apalutamide, participants also undergo stereotactic body radiation therapy for 1-5 fractions.

After completion of study treatment, participants are followed at for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Progressive, castration-resistant prostate cancer demonstrated during continuous antiandrogen therapy (ADT), defined as 3 PSA rises at least 1 week apart, with a minimum PSA > .05 ng/mL obtained during screening.
* At least one but no more than 5 discrete PSMA-avid radiation fields on baseline PSMA-PET scan; all PSMA-avid lesions in radiation fields must be amenable to SBRT in judgment of treating radiation oncologist; there are no restrictions on site of lesion/radiation fields (e.g. bone, lymph node, prostate, visceral). Equivocal lesions/radiation fields on PSMA PET scan that are not definitive for metastasis will not count towards the limit of 5 radiation fields and will not undergo SBRT
* Surgically or medically castrated, with testosterone levels of < 50 ng/dL during screening; if the patient is medically castrated, continuous dosing with luteinizing hormone-releasing hormone (LHRH) analogue must have been initiated at least 4 weeks prior to randomization and must be continued throughout the study to maintain castrate levels of testosterone including post-treatment follow up period
* No prior systemic treatment initiated for the treatment of castration resistant prostate cancer, including abiraterone acetate, enzalutamide, apalutamide, darolutamide, other novel AR or CYP17 antagonist, or docetaxel.
* Patients receiving bone loss prevention treatment with bone-modifying agents (e.g. denosumab, zoledronic acid) must be on stable doses for at least 4 weeks prior to randomization
* Patients who received a first generation anti-androgen (e.g., bicalutamide, flutamide, nilutamide) as most recent treatment must have at least a 6-week washout prior to randomization and must show continuing disease (PSA) progression (an increase in PSA) after washout
* At least 4 weeks or 5 half-lives, whichever is shorter, must have elapsed from the use of any anti-cancer therapy, other than Luteinizing hormone-releasing hormone (LHRH) analog or first generation antiandrogen, prior to randomization
* At least 4 weeks must have elapsed from major surgery or radiation therapy prior to randomization
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status grade 0 or 1
* Resolution of all acute toxic effects of prior therapy or surgical procedure to grade 1 or baseline prior to randomization
* Serum aspartate transaminase (AST) ((serum glutamic oxaloacetic transaminase (SGOT])) and serum alanine transaminase (ALT) (( serum glutamic pyruvic transaminase (SGPT)) ≤ 2.5 x upper limit of normal (ULN)
* Total serum bilirubin ≤ 1.5 x ULN; in subjects with known or suspected Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, direct bilirubin is ≤ 1.5 x ULN
* Glomerular filtration rate ≥ 45 ml/min based on Cockcroft-Gault equation
* Absolute neutrophil count (ANC) ≥ 1500/microliter
* Platelets ≥ 75,000/microliter without transfusion and/or growth factors in the 3 months prior to randomization
* Hemoglobin ≥ 9.0 g/dL without transfusion and/or growth factors in the 3 months prior to randomization
* Serum albumin ≥ 3.0 g/dL
* Signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial prior to randomization
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, and other study procedures, including ability to swallow study drug tablets and long-term follow-up
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug; must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Presence of visceral lesions (e.g. lung, liver) detectable on baseline imaging or bone lesions requiring focal radiation treatment at the time of study entry
* History of seizure or condition that may pre-dispose to seizure (e.g., prior stroke within 1 year prior to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system (CNS) or meningeal disease which may require treatment with surgery or radiation therapy
* Concurrent therapy with any of the following (all must have been discontinued or substituted for at least 1 week prior to randomization, except for medications known to lower seizure threshold which must be discontinued or substituted at least 4 weeks prior to randomization)
* Medications known to lower the seizure threshold
* Herbal (e.g., saw palmetto) and non-herbal (e.g., pomegranate) products that may decrease PSA levels
* Systemic (oral/intravenous (IV)/intramuscular (IM)) corticosteroids; patients on chronic stable dose of steroids at an equivalent dose of prednisone ≤ 10 mg daily may be permitted to enroll at the discretion of principal investigator
* Any other experimental treatment on another clinical trial
* Any of the following within 6 months prior to randomization: Severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias
* Uncontrolled hypertension at study entry; patients with a history of uncontrolled hypertension are allowed provided blood pressure is controlled by antihypertensive treatment
* Gastrointestinal disorder affecting absorption
* Secondary malignancy requiring active treatment except for non-melanoma skin cancer and superficial bladder cancer
* Any medical condition that would be a contra-indication to radiation therapy, such as inflammatory bowel disease
* Spinal cord compression or impending spinal cord compression
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Apalutamide Montherapy): Participants receive apalutamide PO QD on days 1-28. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
- Arm B (Apalutamide, SBRT): Participants receive apalutamide orally (PO) once a day (QD) on days 1-28. Courses repeat every 28 days for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Beginning 60 days after first dose of apalutamide, participants also undergo stereotactic body radiation therapy for 1-5 fractions.
Period: Overall Study
Arm/Group | Arm A (Apalutamide Montherapy) | Arm B (Apalutamide, SBRT)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Apalutamide Monotherapy) | Arm B (Apalutamide, SBRT) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 0 | 1 | 1
  60-69 years old | 2 | 3 | 5
  70-79 years old | 9 | 8 | 17
  80-89 years old | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Undetectable Serum Prostate-specific Antigen (PSA)
Description: The primary endpoint for the study is the proportion of participants with undetectable serum PSA (< 0.2 ng/mL) at 6 months following completion of apalutamide therapy (18 months from date of randomization). Participants who discontinue apalutamide prior to completion of 12 months of therapy for reasons other than disease progression by Prostate Cancer Clinical Trials Working Group (PCWG) criteria, as well as participants who withdraw or are lost to follow up, will be considered unevaluable for this analysis. Participants who discontinue treatment for radiographic or clinical progression, even if occurring prior to receipt of Stereotactic radiation therapy (SBRT) in the experimental arm), would be evaluable for analysis of the primary endpoint.
Time Frame: Approximately 18 months from date of randomization
Measure: Number; unit: proportion of participants
Arm/Group | Arm A (Apalutamide Monotherapy) | Arm B (Apalutamide, SBRT)
Number analyzed (Participants) | 13 | 13
proportion of participants | 0 | 0.308

2. Secondary Outcome: Median Time to PSA Progression
Description: Time to a diagnosis of PSA progression defined by the Prostate Cancer Working Group (PCWG) criteria will be estimated using Kaplan-Meier methods for each treatment arm and will be used to estimate the median time to progression and 95% confidence interval (CI).
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Apalutamide Montherapy) | Arm B (Apalutamide, SBRT)
Number analyzed (Participants) | 13 | 13
months | 13.82 [9.21 to NA] — There were insufficient number of events so an upper limit to for the confidence interval could not be calculated. | NA [30.16 to NA] — There were insufficient number of events, so a median and confidence interval could not be calculated.

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events (AEs)
Description: For each treatment arm, adverse event incidence per group will be summarized by severity (highest grade) for those AEs judged by the Investigator to be probably, possibly, or definitely related to the study treatment and will be summarized by frequency and percentage, with all participants treated in that treatment arm as the denominator unless otherwise specified. In addition, Adverse events with missing severity or relationship to study drug will be classified as severe and treatment-related, respectively.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Apalutamide Monotherapy) | Arm B (Apalutamide, SBRT)
Number analyzed (Participants) | 13 | 13
Participants
  Alopecia, Grade 1 | 0 | 1
  Blurred Vision, Grade 1 | 0 | 1
  Constipation, Grade 1 | 1 | 1
  Depression, Grade 1 | 0 | 2
  Diarrhea, Grade 2 | 0 | 1
  Dizziness, Grade 1 | 1 | 2
  Dysgeusia, Grade 1 | 1 | 0
  Fatigue, Grade 3 | 1 | 0
  Hallucinations, Grade 1 | 0 | 1
  Hot Flashes, Grade 3 | 1 | 0
  Hypertension, Grade 3 | 0 | 1
  Hypothyroidism, Grade 2 | 2 | 0
  Lymphocyte count decreased, Grade 3 | 0 | 2
  Muscle weakness lower limb, Grade 1 | 1 | 0
  Nausea, Grade 1 | 1 | 1
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify, Grade 1 | 1 | 1
  Neutrophil count decreased, Grade 2 | 0 | 1
  Pruritus, Grade 2 | 0 | 1
  Rash maculo-papular, Grade 3 | 0 | 1
  White blood cell decreased, Grade 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | Arm A (Apalutamide Monotherapy) | Arm B (Apalutamide, SBRT)
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Apalutamide Monotherapy) (N=13) | Arm B (Apalutamide, SBRT) (N=13)
Hematuria (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Apalutamide Monotherapy) (N=13) | Arm B (Apalutamide, SBRT) (N=13)
Hypothyroidism (Endocrine disorders) | 3 (5) | 1 (1)
Eye Disorders - Other, specify (Eye disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (7)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 8 (11) | 10 (13)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1)
Eye Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (11)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot Flashes (Vascular disorders) | 3 (4) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03503344/Prot_SAP_000.pdf